CLINICAL TRIAL: NCT06114199
Title: Enhancing the Effectiveness of Home-delivery Based Produce Prescription Program Implementation Strategies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Nalini Ranjit, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-23-0734 (substudy)
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Nutritional Deficiency in Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Produce Prescription Program (PPRx) Standard (Active Comparator): Participants will receive biweekly deliveries of 20 lbs (~50 servings) of fresh produce (8-10 different kinds of produce) plus standard nutrition education materials consisting of nutrition education infographics inside of the produce prescription boxes as well as online videos, recipes, and nutrition tips accessed via Quick Response (QR) code.
  Interventions: Behavioral: Produce Prescription Program (PPRx) Standard
- Produce Prescription Program (PPRx) Standard plus Smartphone App (Experimental): Participants will receive biweekly deliveries of 20 lbs (~50 servings) of fresh produce (8-10 different kinds of produce) plus the same standard nutrition education materials provided to the control group consisting of nutrition education infographics inside of the produce prescription boxes as well as online videos, recipes, and nutrition tips accessed via Quick Response (QR) code. Additionally, participants will be given access to a smartphone app that allows women to interact with an artificial intelligence (AI) chatbot to obtain real-time cooking suggestions.
  Interventions: Behavioral: Produce Prescription Program (PPRx) Standard; Behavioral: Smartphone App

INTERVENTIONS:
Behavioral: Produce Prescription Program (PPRx) Standard — Participants will receive biweekly deliveries of 20 lbs (~50 servings) of fresh produce (8-10 different kinds of produce) plus standard nutrition education materials consisting of nutrition education infographics inside of the produce prescription boxes as well as online videos, recipes, and nutrition tips accessed via Quick Response (QR) code.
Behavioral: Smartphone App — Participants will be given access to a smartphone app that allows women to interact with an artificial intelligence (AI) chatbot to obtain real-time cooking suggestions.
  Arms: Produce Prescription Program (PPRx) Standard plus Smartphone App

SUMMARY:
Harris Health System is currently participating, along with two other partners, GoldiFresh Inc., and Brighter Bites, in a cross-sector collaborative home delivery-based Produce Prescription Program (PPRx) pilot initiative that provides consistent access to healthy food plus nutrition education to Medicaid-eligible pregnant women in Harris County, TX, deemed to be at high risk of adverse pregnancy or birth outcomes. The objectives of this study are two-fold: (a) to examine utilization of food basket contents and improvements in diet quality in this home delivery based PPRx program, and (b) to evaluate if and the extent to which utilization of food basket contents outcomes improves with support from an interactive AI-based conversational agent to convert food into healthy meals.

ELIGIBILITY:
Inclusion Criteria:

* receiving prenatal care at high-risk obstetric clinics
* <= 20 weeks medically-confirmed viable pregnancy
* designated as high risk [Age>=35 years, or obese or overweight (BMI>=25.0 at pre pregnancy self-report), or prior history of pregnancy hypertension or gestational diabetes]
* within the zip code delivery radius

Exclusion Criteria:

* women who were medically recommended bed rest through pregnancy
* substance users

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Change in consumption of home-delivered produce from baseline to 6 months | Measures will be collected at baseline, and 6 times at random intervals over the next 6 months
  7 point rating scale ranging from 0=none to 6=all, assessing what proportion of delivered produce was consumed over the past two weeks.
Change in usual consumption of fruits and vegetables from baseline to 6 months | Measures will be collected at baseline, and after 6 months of exposure to program
  Fruit and vegetable consumption scale, measured by NCI dietary screener. Scale includes multiple sources of fruit and vegetables in diet, and is scored in terms of cups of fruit / day, and cups of vegetables / day

CONTACTS AND LOCATIONS:
Overall Officials: Nanlini Ranjit, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
At the end of the project, de-identified data at individual level will be uploaded to the American Heart Association (AHA) Precision-Medicine Platform.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: September 30, 2024
Access Criteria: Will be determined by AHA.